CLINICAL TRIAL: NCT06168721
Title: Development of an ICF Core Set for the Management of Musculoskeletal Conditions in Primary Care Physiotherapy Services
Brief Title: ICF Core Set for Primary Care Physiotherapy
Status: Completed | Type: Observational
Sponsor: University of Valladolid (Other)
Collaborators: Sanidad de Castilla y León (Other)
Responsible Party: Principal Investigator, Héctor Hernández Lázaro, Adjunct Professor, University of Valladolid
Other Study IDs: CEIm 2987
Record Dates: First submitted 2023-12-04; First posted 2023-12-13 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Musculoskeletal Diseases
Keywords: ICF; Musculoskeletal Diseases; Physical Therapy Modalities; Primary Health Care; Community Health Services
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Expert panel: This group will be composed of experts in primary care physiotherapy.
  Interventions: Other: Expert survey

INTERVENTIONS:
Other: Expert survey — The expert group will participate in a two-round survey using the Delphi method. The first round aims to assess the relevance of the proposed ICF categories and to identify missing concepts. The second round will aim to confirm the appropriateness of including the selected categories in the ICF core set. Each round will last 3 weeks and the experts will be provided with feedback on the results obtained.

SUMMARY:
Primary care physiotherapy services provide community-based care for musculoskeletal conditions. These conditions are often associated with disability and impact on patients' quality of life. The International Classification of Functioning, Disability and Health (ICF) is the global framework for describing disability. ICF Core Sets are ICF-based tools that facilitate the clinical use of this classification. The development of these tools follows a scientific process that combines the perspectives of researchers, patients, professionals, and the care setting. Our research team has conducted preliminary studies and identified candidate ICF categories with good potential for inclusion in a preliminary version of an ICF Core Set for the treatment of musculoskeletal conditions in community physical therapy settings. The aim of this study is to confirm the relevance of the candidate categories and to develop a final version of this ICF Core Set.

DETAILED DESCRIPTION:
Primary care physiotherapy services provide community-based care for musculoskeletal conditions. These conditions are often associated with disability and impact on patients' quality of life. The International Classification of Functioning, Disability and Health (ICF) is the global framework for describing disability. ICF Core Sets are ICF-based tools that facilitate the clinical use of this classification. Some ICF Core Sets are designed to describe the functioning of patients with musculoskeletal problems.

These Core Sets are focused on the acute phase, typical of emergency care, and the post-acute phase, intended for multidisciplinary teams in rehabilitation centers. However, no ICF core set exists for the final stages of these conditions, when the patient has been reintegrated into the community. The development of ICF Core Sets follows a scientific process that integrates the perspectives of researchers, patients, professionals, and the care setting. Therefore, preparatory studies have been carried out, taking as a reference the physiotherapy services in primary care, where most of these conditions are treated.

These preparatory studies have made it possible to draw up a list of ICF categories that are candidates for being part of an ICF core set specific to these services. To confirm the relevance of these categories, a cross-sectional observational study will be developed by recruiting a group of experts. The experts will carry out two rounds of the survey according to the Delphi method. To be part of this group, sufficient expertise in the field of primary care physiotherapy will be required. The categories that reach consensus among these experts will be proposed in the development of a tailored ICF Core Set for primary care physiotherapy services.

The aim of this study is to confirm the relevance of the candidate categories and to develop a final version of an ICF Core Set for the management of musculoskeletal conditions in a primary care physiotherapy clinical setting. The availability of this tool would allow guiding physical therapy assessments, selecting optimal outcome measures, implementing person-centered care, and systematically recording clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Be physiotherapists working in a primary care setting for the duration of the study.
* Have more than 5 years of experience in this clinical setting.
* Evidence of completion of at least 200 hours of additional training, teaching, research, and/or administrative activities related to the clinical setting.

Exclusion Criteria:

* Work in a rehabilitation center or hospital context.

Ages: 26 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The potential participants in this study should be physical therapists working in a primary care clinical setting. The resulting panel of experts would have sufficient expertise in this area. The study will focus on the Spanish region of 'Castilla and Leon', but efforts will be made to extend the scope to a national level.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
Relevance of candidate ICF categories (First Delphi Round) | 2024-01/2024-06
  The relevance of the categories will be measured on a 5-point Likert scale: "not relevant" (score 1), "hardly relevant" (score 2), "somewhat relevant" (score 3), "relevant" (score 4) and "very relevant" (score 5).
Judgment on the clinical utility of the selected ICF categories (Second Delphi Round) | 2024-01/2024-06
  Dichotomous question (yes/no) on the appropriateness of including or excluding the most relevant ICF categories in the ICF core set.

SECONDARY OUTCOMES:
Missing functioning concepts (First Delphi Round) | 2024-01/2024-06
  Open-ended question related to ICF

OTHER OUTCOMES:
Sociodemographic data of the sample | 2024-01/2024-06
  Data set for the characterization of the expert panel (age, gender, education level, work experience and information on the current job)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Jiménez del Barrio, PhD, Study Chair — University of Valladolid; Luis Ceballos Laita, PhD, Study Chair — University of Valladolid; María Teresa Mingo Gómez, PhD, Study Chair — University of Valladolid
Locations (1):
- Ólvega Primary Health Center, Ólvega, Soria, Spain

IPD SHARING:
Plan to Share IPD: Yes
The authors confirm that the data supporting the findings of this study will be available within the article and/or its supplementary materials.
Supporting Information: Study Protocol, SAP
Time Frame: From the publication of the study, with no time limit.
Access Criteria: Access to this data will be conditioned by the type of publication.

REFERENCES:
- [Background] Hernandez-Lazaro H, Mingo-Gomez MT, Ceballos-Laita L, Medrano-de-la-Fuente R, Jimenez-Del Barrio S. Validation of the international classification of functioning, disability, and health (ICF) core sets for musculoskeletal conditions in a primary health care setting from physiotherapists' perspective using the Delphi method. Disabil Rehabil. 2023 Jul;45(15):2458-2468. doi: 10.1080/09638288.2022.2096128. Epub 2022 Jul 13. PMID 35830343
- [Background] Hernandez-Lazaro H, Mingo-Gomez MT, Jimenez-Del-Barrio S, Lahuerta-Martin S, Hernando-Garijo I, Medrano-de-la-Fuente R, Ceballos-Laita L. Researcher's Perspective on Musculoskeletal Conditions in Primary Care Physiotherapy Units through the International Classification of Functioning, Disability, and Health (ICF): A Scoping Review. Biomedicines. 2023 Jan 20;11(2):290. doi: 10.3390/biomedicines11020290. PMID 36830831
- [Background] Hernandez-Lazaro H, Mingo-Gomez MT, Jimenez-Del-Barrio S, Rodriguez-Fernandez AI, Areso-Boveda PB, Ceballos-Laita L. Validation of the International Classification of Functioning, Disability, and Health (ICF) core set for post-acute musculoskeletal conditions in a primary care physiotherapy setting from the perspective of patients using focus groups. Disabil Rehabil. 2024 Aug;46(16):3594-3601. doi: 10.1080/09638288.2023.2251392. Epub 2023 Sep 5. PMID 37667886
- [Background] Hernandez-Lazaro H, Jimenez-Del Barrio S, Ceballos-Laita L, Lahuerta-Martin S, Medrano-de-la-Fuente R, Hernando-Garijo I, Mingo-Gomez MT. Multicentre cross-sectional study assessing content validity of the International Classification of Functioning, disability and health core set for post-acute musculoskeletal conditions in primary care physiotherapy services. J Rehabil Med. 2023 Nov 16;55:jrm11950. doi: 10.2340/jrm.v55.11950. PMID 37974517
- [Result] Hernandez-Lazaro H, Mingo-Gomez MT, Jimenez-Del-Barrio S, Simarro-Martin A, Wisniowska-Szurlej A, Ceballos-Laita L. Development of an ICF core set for the management of musculoskeletal conditions in primary care physiotherapy services in Spain: a Delphi study. Disabil Rehabil. 2025 Sep;47(18):4759-4768. doi: 10.1080/09638288.2025.2460723. Epub 2025 Feb 11. PMID 39931756